CLINICAL TRIAL: NCT01943565
Title: Intrathecal Hydromorphone for Post-cesarean Delivery Pain - a Dose Finding Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Research question answered by another group of researchers (Sviggum et al)
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Dirk Varelmann, MD, Instructor of Anaesthesiology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2013P001850; Hydromorphone_IT (Other: BrighamHospital)
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-05

CONDITIONS: Healthy; Pain; Pregnancy
Keywords: Pregnancy; Healthy; Intrathecal; Opioids; Spinal; Anesthesia; Pain; Cesarean; Delivery; Human
MeSH Terms: conditions — Pain | interventions — Hydromorphone; Anesthesia, Spinal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hydromorphone 25mcg (Active Comparator): The arm will receive 25mcg intrathecal hydromorphone to supplement the spinal anesthesia
  Interventions: Drug: Hydromorphone 25mcg; Drug: spinal anesthesia
- Hydromorphone 50mcg (Active Comparator): The arm will receive 50mcg intrathecal hydromorphone to supplement the spinal anesthesia
  Interventions: Drug: Hydromorphone 50mcg; Drug: spinal anesthesia
- Hydromorphone 100mcg (Active Comparator): The arm will receive 100mcg intrathecal hydromorphone to supplement the spinal anesthesia
  Interventions: Drug: Hydromorphone 100mcg; Drug: spinal anesthesia

INTERVENTIONS:
Drug: Hydromorphone 25mcg — Intrathecal Hydromorphone 25mcg
  Other Names: HM25
  Arms: Hydromorphone 25mcg
Drug: Hydromorphone 50mcg — Intrathecal Hydromorphone 50mcg
  Other Names: HM50
  Arms: Hydromorphone 50mcg
Drug: Hydromorphone 100mcg — Intrathecal Hydromorphone 100mcg
  Other Names: HM100
  Arms: Hydromorphone 100mcg
Drug: spinal anesthesia — bupivacaine 0.75% 1.6 mL (12mg)

SUMMARY:
Pain relief after cesarean delivery can be provided in a few ways. Most commonly, certain medications called opioids, such as morphine, are given through the vein or into the muscle. However, a more effective way to give pain relief with fewer side effects (such as nausea and slowing your breathing) is to give opioids in the spinal space as part of the medications given for a cesarean delivery.

For many years, the opioid of choice was morphine due to its long anesthetic effect and acceptable side effect profile. A nation-wide disruption in the supply of preservative-free morphine has made it necessary to look for alternatives. Many institutions worldwide have used another opioid, called hydromorphone, in the spinal space for over a decade. This drug has a very good safety and side effect profile and has been used at the investigators' institution for more than a year. Of interest, while a number of different doses of hydromorphone have been used, there have been very few studies to evaluate the best dose for providing good pain relief with minimal side effects. The goal of this study is to find the best dose of spinal hydromorphone for women undergoing cesarean delivery.

DETAILED DESCRIPTION:
Intrathecal opioids in have been shown to produce analgesia. Lipid solubility and effect on specific mu opioid receptors in the dorsal horn of the spinal cord primarily determine the analgesic effect of intrathecally injected opioids. Rostral spread of intrathecal opioids causes some of the side effects like pruritus, respiratory depression, nausea and vomiting.

In the investigators' institute, during cesarean delivery under spinal anesthesia is usually performed with 1.6-1.8 ml of 0.75% bupivacaine with dextrose (hyperbaric solution) with 10-20mcg of fentanyl. Preservative free intrathecal (IT) morphine100 to 200 mcg is injected at the time of initiation of spinal block for postoperative pain relief. Multiple studies have shown excellent postoperative pain relief following cesarean delivery up to 18hrs with this dosing regimen.

However, there has been a national shortage of preservative free morphine since August 2012. Based on the pharmacokinetic and pharmacodynamic profile, intrathecal (IT) preservative free hydromorphone 100 mcg has been used as a substitute. Anecdotal experience during the past 8 months suggest that patients have comparable post partum pain relief, with a similar side-effect profile to IT morphine.

There is no published data on the optimal dose of IT hydromorphone for post cesarean analgesia. There are case reports and retrospective case study of use of 100mcg IT hydromorphone. One randomized controlled trial for knee arthroscopy used 2.5-5-10 mcg of IT hydromorphone for postoperative analgesia.

Hence it is important to determine the optimal dose of IT hydromorphone for post operative pain management following cesarean delivery in terms of analgesic efficacy, incidence of side effects and the need for treatment interventions

This study will aim to determine the optimal dose of intrathecal hydromorphone that would provide adequate postoperative analgesia with minimal side effects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy at-term parturients undergoing elective cesarean delivery under spinal anesthesia

Exclusion Criteria:

* Emergency cesarean delivery
* Respiratory disease
* significant comorbidities: preeclampsia, insulin-dependent diabetes mellitus
* obstructive sleep apnea
* body mass index > 35kg/m2
* <18yrs
* documented intolerance or allergy to systemic or neuraxial opioids
* patient with a history of chronic opioid or current use of opioids

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk J Varelmann, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Wang JK, Nauss LA, Thomas JE. Pain relief by intrathecally applied morphine in man. Anesthesiology. 1979 Feb;50(2):149-51. doi: 10.1097/00000542-197902000-00013. No abstract available. PMID 373503
- [Background] Ross BK, Hughes SC. Epidural and spinal narcotic analgesia. Clin Obstet Gynecol. 1987 Sep;30(3):552-65. doi: 10.1097/00003081-198709000-00010. No abstract available. PMID 2888557
- [Background] Palmer CM, Emerson S, Volgoropolous D, Alves D. Dose-response relationship of intrathecal morphine for postcesarean analgesia. Anesthesiology. 1999 Feb;90(2):437-44. doi: 10.1097/00000542-199902000-00018. PMID 9952150
- [Background] Milner AR, Bogod DG, Harwood RJ. Intrathecal administration of morphine for elective Caesarean section. A comparison between 0.1 mg and 0.2 mg. Anaesthesia. 1996 Sep;51(9):871-3. doi: 10.1111/j.1365-2044.1996.tb12622.x. PMID 8882255
- [Background] Lee YS, Park YC, Kim JH, Kim WY, Yoon SZ, Moon MG, Min TJ. Intrathecal hydromorphone added to hyperbaric bupivacaine for postoperative pain relief after knee arthroscopic surgery: a prospective, randomised, controlled trial. Eur J Anaesthesiol. 2012 Jan;29(1):17-21. doi: 10.1097/EJA.0b013e3283476055. PMID 21562420

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydromorphone 25mcg | Hydromorphone 50mcg | Hydromorphone 100mcg
Started | 11 | 9 | 9
Completed | 11 | 9 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydromorphone 25mcg | Hydromorphone 50mcg | Hydromorphone 100mcg | Total
Number analyzed (Participants) | 11 | 9 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 10 | 30
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 10 | 30
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 9 | 10 | 30

OUTCOME MEASURES:

1. Primary Outcome: 24hr Post-partum IV Opioid Requirement
Description: Intrathecal (IT) hydromorphone added to intrathecally administered local anesthetics for spinal anesthesia increases patient comfort by decreasing post-operative pain. This leads to a decrease in the post-operative intravenous hydromorphone requirements.
Time Frame: 24hrs after administration of intrathecal hydromorphone
Population: One 25 mcg patient is missing data on this outcome
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Hydromorphone 25mcg | Hydromorphone 50mcg | Hydromorphone 100mcg
Number analyzed (Participants) | 10 | 9 | 9
mg | 3.44 (3.51) | 3.11 (2.15) | 4.40 (3.51)

2. Secondary Outcome: Oxygen Saturation, Need for Supplemental Oxygen
Description: Intravenously, and to a lesser extent, intrathecally administered opioids can lead to respiratory depressions. Therefore the subjects' oxygen saturation is measured (standard clinical practice).
Time Frame: 24hrs post administration of IT hydromorphone
Population: One 25 mcg patient is missing data on this outcome
Measure: Mean (Standard Deviation); unit: percentage oxygenated haemoglobin
Arm/Group | Hydromorphone 25mcg | Hydromorphone 50mcg | Hydromorphone 100mcg
Number analyzed (Participants) | 10 | 9 | 9
percentage oxygenated haemoglobin | 98.3 (1.49) | 99.0 (0.87) | 98.4 (1.33)

3. Secondary Outcome: Patients With Nausea and Vomiting Requiring Rescue Medication
Description: IV and IT opioids can induce nausea and vomiting. Outcome measure is reported as percentage of patients with nausea and vomiting requiring rescue medication.
Time Frame: 24hrs post administration of IT hydromorphone
Population: One 25 mcg patient was missing data on this measure
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone 25mcg | Hydromorphone 50mcg | Hydromorphone 100mcg
Number analyzed (Participants) | 10 | 9 | 9
Participants | 3 | 2 | 2

4. Secondary Outcome: Number of Patients With Hypothermia (Body Temperature < 95F/35C)
Description: intrathecally administered opioids can cause hypothermia (body temperature <95F/35C)
Time Frame: 24hrs post administration of IT hydromorphone
Population: One 25 mcg patient was missing data on this measure
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone 25mcg | Hydromorphone 50mcg | Hydromorphone 100mcg
Number analyzed (Participants) | 10 | 9 | 9
Participants | 0 | 0 | 0

5. Secondary Outcome: Number of Patients With Visual Disturbances
Description: IT/IV opioids can create visual disturbances. The number of patients with visual disturbances are reported.
Time Frame: 24hrs post administration of IT hydromorphone
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone 25mcg | Hydromorphone 50mcg | Hydromorphone 100mcg
Number analyzed (Participants) | 11 | 9 | 9
Participants | 0 | 0 | 0

6. Secondary Outcome: Number of Patients With Pruritus
Description: IT opioids can cause pruritus. Persistent pruritus requiring treatment will be recorded.
Time Frame: 24hrs post administration of IT hydromorphone
Population: One 25 mcg patient is missing data on this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Hydromorphone 25mcg | Hydromorphone 50mcg | Hydromorphone 100mcg
Number analyzed (Participants) | 10 | 9 | 9
Participants | 0 | 4 | 3

7. Secondary Outcome: Intraoperative Vasopressor Use: Ephedrine Equivalents
Description: IT (intrathecal) applied local anesthetics and opioids can cause arterial and venous vasodilation leading to a decrease in afterload as well as preload. This is typically treated with volume replacement and vasopressors (acutely). Total intraoperative vasopressor use will be reported for ephedrine equivalents.
Time Frame: Intraoperatively (at time of operation)
Population: One 25 mcg patient is missing data on this outcome
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Hydromorphone 25mcg | Hydromorphone 50mcg | Hydromorphone 100mcg
Number analyzed (Participants) | 10 | 9 | 9
mg | 60.98 (26.94) | 56.48 (32.27) | 45.48 (19.78)

8. Secondary Outcome: Intraoperative Vasopressor Use: Phenylephrine Equivalents
Description: IT (intrathecal ) applied local anesthetics and opioids can cause arterial and venous vasodilation leading to a decrease in afterload as well as preload. This is typically treated with volume replacement and vasopressors (acutely).
  Total intraoperative vasopressor use will be reported for phenylephrine equivalents.
Time Frame: Intraoperatively (at time of operation)
Population: One 25 mcg patient is missing data on this outcome
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Hydromorphone 25mcg | Hydromorphone 50mcg | Hydromorphone 100mcg
Number analyzed (Participants) | 10 | 9 | 9
mcg | 751.04 (331.76) | 695.54 (397.42) | 560.11 (243.56)

ADVERSE EVENTS:
Arm/Group | Hydromorphone 25mcg | Hydromorphone 50mcg | Hydromorphone 100mcg
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 1/11 | 1/9 | 1/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydromorphone 25mcg (N=11) | Hydromorphone 50mcg (N=9) | Hydromorphone 100mcg (N=9)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes